CLINICAL TRIAL: NCT00432263
Title: Placebo-Controlled Trial On The Efficacy Of Growth Hormone Replacement Therapy In Patients With Growth Hormone Deficiency After Traumatic Brain Injury
Brief Title: Treatment Of Adult Growth Hormone Deficiency After Traumatic Brain Injury.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6281274
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Human Growth Hormone

INTERVENTIONS:
Drug: Genotropin (PN-180,307) Somatropin

SUMMARY:
To establish the effects of genotropin replacement in patients with severe growth hormone deficiency after traumatic brain injury on cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Have had a previous traumatic brain injury (more than 1 year and less than 5 years) prior to the screening visit.
* Have an Extended Glasgow Outcome Scale (GOS-E) more than or equal to 5.

Exclusion Criteria:

* Active systemic malignancy or active intracranial tumor. A successfully treated tumor or malignancy is not an exclusion criterion if the patient has not had active disease for 5 years and is not currently receiving maintenance chemotherapy, (except for basal cell skin cancers.
* Receiving treatment with prednisolone in doses above 10 mg/day or treatment with other oral glucocorticosteroids above replacement doses is not permitted throughout the study. Topical and inhaled corticosteroids are permitted.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-04

PRIMARY OUTCOMES:
The primary endpoint is the change from baseline in the CogState™ composite score at Week 36.

SECONDARY OUTCOMES:
Change CogState™ at Week 12, 24, 60 and 72. Change in lean body mass and fat mass at Week 36 and 72. Change in the Extended Glasgow Outcome Scale at week 36 and 72. Change in quality of life at week 24, 36, 60 and 72. Summary of change in cardiovascular

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281274&StudyName=Treatment+Of+Adult+Growth+Hormone+Deficiency+After+Traumatic+Brain+Injury%2E